CLINICAL TRIAL: NCT04554095
Title: Development of a Multimodal Index to Improve the Predictive Value of Success in Weaning From Mechanical Ventilation
Status: Recruiting | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Candelaria de Haro, Medical doctor and Doctor of Philosophy, Corporacion Parc Tauli
Other Study IDs: Multimodal Weaning
Record Dates: First submitted 2020-08-31; First posted 2020-09-18 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Weaning Failure; Mechanical Ventilation Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Clinical data collection — Respiratory parameters, analytic values, lung ultrasound and echocardiography

SUMMARY:
Weaning from mechanical ventilation (MV) is a complex process in which patients are liberated from the ventilator. Prolongued weaning and weaning failure, defined as the need for reintubation, have different adverse effects, including prolongation of MV, intensive care unit (ICU) and hospital stay, and are also associated with increased incidence of ventilator-associated pneumonia and high mortality. The rate of weaning failure is high, even when the classic extubation criteria are met, so it is necessary to improve scores that allow predicting and determining the ideal time for MV withdrawal.

The aim of this study is to design a new multimodal index to predict and optimize weaning results in a personalized way, based on the use and interpretation of data derived from continuous monitoring of critically ill patients. The new multimodal index, in addition to classical respiratory parameters, will include parameters related to patient-ventilator interaction (asynchronies), diaphragmatic function, cardiovascular status and autonomic nervous system function (ANS).

The investigators have designed a prospective observational study that will include 126 critical patients from a medical-surgical ICU that meet the classical criteria for weaning. The management of the patients, as well as the weaning process, will be carried out following the usual protocol. In addition to the classical weaning predictor data, data on the patient-ventilator interaction and the function of the autonomic nervous system will be collected by means of specific software (BetterCare). Cardiovascular and diaphragmatic function will be evaluated using ultrasound. Based on the advanced analysis of data from different devices collected throughout the mechanical ventilation period, it will be designed a "personalized" weaning score that should improve the accuracy of the decision-making process and therefore reduce morbidity and mortality. Additional benefits would include lowering health care costs without increasing adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MV> 24 hours.
* Patients with orotracheal tube.
* Patients who meet the classic criteria of weaning from the MV defined as:

Improvement or resolution of the cause required for MV. PaO2> 60mmHg with FiO2≤0.4 and PEEP ≤8cm H2O. Glasgow Coma Score> 10 Temperature <38 ° C. Hemoglobin> 8g / dL No need for vasoactive drugs or at doses <5μg / kg / min Obtaining informed consent.

Exclusion Criteria:

* Tracheostomy patients.
* Patients with neurological pathology with involvement of the brainstem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU of the Parc Taulí Universitary Hospital undergoing MV and starting the weaning process according to the protocol established for usual clinical care practice.
Sampling Method: Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Multimodal index for weaning prediction evaluation | 48 hours after mechanical ventilation withdrawal
  Number of successful weanings evaluated through the new multi-modal index compared to the classic indexes

SECONDARY OUTCOMES:
Predictive value of patient-ventilator interaction | From day 1 of mechanical ventilation until 48 hours after mechanical ventilation withdrawal
  association between asynchronies and weaning failure

CONTACTS AND LOCATIONS:
Locations (1):
- Candelaria De Haro, Sabadell, Barcelona, Spain